CLINICAL TRIAL: NCT07184268
Title: Clinical Efficacy of Non-surgical Therapy With Local Delivery of Ozonated Olive Oil Gel Versus Curcumin Gel in Stage II Grade B Periodontitis Randomized Controlled Clinical Trial.
Brief Title: Clinical Efficacy of NST With Local Delivery of Ozonated Olive Versus Curcumin Gel in Stage II Grade B Periodontitis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: MTI University (Other)
Responsible Party: Principal Investigator, Parryhan Mohamed Abdelsamie, Lecturer of periodontology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 892025
Record Dates: First submitted 2025-09-08; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Periodontitis, Adult
Keywords: Nonsurgical therapy; local delivery gel; curcumin gel; ozonated olive oil; molar incisor pattern periodontitis; Chronic periodontitis; stage II grade B
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Intervention Model Description: The test group "Group 1" will receive full Scaling and root planing (SRP) followed by subgingival application of ozonated olive gel.
  The control group "Group 2" will receive full-mouth SRP followed by subgingival application of curcumin gel
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- curcumin gel (Active Comparator): The curcumin gel will be gently deposited into the periodontal pockets to ensure adequate subgingival delivery.
  Interventions: Procedure: full mouth non-surgical scaling
- ozonated olive gel. (Active Comparator): patients will receive subgingival application of ozonated olive oil in the periodontal pocket
  Interventions: Procedure: full mouth non-surgical scaling

INTERVENTIONS:
Procedure: full mouth non-surgical scaling — All patients will receive a full mouth scaling using ultrasonic scalers and hand instrumentation

SUMMARY:
The aim of this clinical trial is to evaluate the effectiveness of local delivery ozonated olive gel versus curcumin gel as adjunct to scaling and root planing in the treatment of stage II grade B periodontitis in on both males and females in the age group between 18 and 50 years. outcome measures are Clinical attachment level (CAL), plaque index (PI), gingival index (GI).

DETAILED DESCRIPTION:
Periodontitis is an advanced periodontal disease with a distinctive clinical signs and symptoms as rapid attachment loss and bone destruction

The primary treatment approach for periodontitis is mechanical plaque removal through debridement, particularly scaling and root planing (SRP) using hand or ultrasonic instruments.

curcumin gel is an adjunct to non-surgical periodontal therapy is a highly potent local antioxidant and anti-inflammatory agent. While ozone has a potent antimicrobial and anti-inflammatory effects it also can be incorporated into a lipid carrier such as olive oil. Ozone's stability and ease of application are markedly enhanced. Ozonized olive oil can be formulated into a gel with ideal rheological properties for injection into periodontal pockets.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with stage II periodontitis defined by having interdental CAL 3-4 mm and presence of pocket depth (PD) ≤ 5 mm, and grade B periodontitis characterized by a moderate rate of disease progression.
2. Patients agree to a 3-month follow-up period and provide an informed consent.

Exclusion Criteria:

1. Presence of prosthetic crowns, overhanging restorations and orthodontic treatment.
2. Teeth with both endo-perio lesions.
3. Antibiotics therapy that has an impact on the clinical signs and symptoms of periodontitis in the previous 3 months.
4. Anti-inflammatory drugs in the previous 1 month.

6. History of systemic disease, allergy, cardiovascular diseases, diabetes mellitus, hypertension, bleeding disorders, hyperparathyroidism, and compromised medical conditions, pregnant and lactating females.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level | 3 months
  measured from the cementoenamel junction (CEJ) to the bottom of pocket.

SECONDARY OUTCOMES:
Gingival Index | 3 months
  Index scores will be recorded showing gingival bleeding and inflammation
Plaque index | 3 months
  be used to evaluate plaque accumulation

CONTACTS AND LOCATIONS:
Overall Officials: Parryhan M Abdelsamie, Principal Investigator — MTI University

IPD SHARING:
Plan to Share IPD: No